CLINICAL TRIAL: NCT06876909
Title: Clinical Effect Observation of Barley Green Intervention in Hyperuricemia Population and Related Mechanism Study of Xanthine Oxidase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Cui Mingxuan, Principal Investigator, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021PHB074-001
Record Dates: First submitted 2025-02-25; First posted 2025-03-14 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-02

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention)
- intervention group (Experimental)
  Interventions: Dietary Supplement: barley green

INTERVENTIONS:
Dietary Supplement: barley green — Oral administration: 30 minutes before meals Dosage: 4 g powder, 5 g tablet Frequency: 2 times a day
  Arms: intervention group

SUMMARY:
This study aims to explore the changes in metabolic-related indicators in patients with hyperuricemia under the intervention of barley green, reveal the clinical effect of barley green in regulating uric acid metabolism, and preliminarily clarify the mechanism of barley green influencing uric acid metabolism through in vitro experiments related to xanthine oxidase. This study plans to recruit patients with hyperuricemia who visit the clinical nutrition department and rheumatology and immunology department of Peking University People's Hospital, randomly dividing them into an intervention group and a control group. The intervention group will take barley green plus a balanced diet plan, while the control group will only be given a balanced diet plan. General clinical data will be collected, and nutritional measurements will be conducted. Venous blood will be drawn for the determination of uric acid metabolism-related indicators, xanthine oxidase activity, and inflammatory factor levels. The differences in uric acid and related metabolic indicators, as well as xanthine oxidase activity, between the two groups will be observed and compared to provide a scientific basis for the clinical application of barley green in non-pharmacological intervention and medical nutrition therapy for hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years old; under a normal purine diet, the fasting blood uric acid level on two different days: 420 μmol/L < blood uric acid < 540 μmol/L (for men), 360 μmol/L < blood uric acid < 540 μmol/L (for women); willing to accept the assessment and sign the informed consent.

Exclusion Criteria:

* ① Patients currently receiving drug treatment for hyperuricemia;

  * Patients with diseases affecting food digestion and absorption (such as chronic diarrhea, constipation, severe digestive tract inflammation, active peptic ulcers, post-gastrointestinal resection, cholecystitis/cholecystectomy, etc.);

    * Patients with cardiovascular and cerebrovascular diseases, grade 3 hypertension, chronic hepatitis, malignant tumors, anemia (hemoglobin value below the normal reference range), mental disorders and memory impairment, epilepsy, etc.;

      * Patients simultaneously receiving other functional food nutritional support (plant active substances, health foods);

        * Patients with abnormal liver function (alanine aminotransferase or/and aspartate aminotransferase exceeding 3 times the upper limit of the normal value); patients with abnormal kidney function (serum creatinine exceeding the upper limit of the normal value);

          * Patients with active pulmonary tuberculosis, AIDS and other infectious diseases; ⑦ Patients with severe allergies to the ingredients of the study nutritional product;

            * Pregnant or lactating women;

              * Patients with limb disabilities and those deemed unsuitable for participation in the study by the clinical doctor (for example, patients with severe diseases not listed in the exclusion criteria); ⑩ Patients with gouty arthritis attacks ≥ 2 times; ⑪ Patients with one gouty arthritis attack and blood uric acid > 480 μmol/L, or combined with any of the following: age < 40 years old, evidence of tophi or urate deposition in the joint cavity, uric acid nephrolithiasis or renal function impairment (eGFR ≤ 89 ml/(min·1.73 m²)), hypertension, impaired glucose tolerance or diabetes, dyslipidemia (any of the four lipid indicators exceeding the normal reference range), obesity (BMI ≥ 28 kg/m²), coronary heart disease, stroke, heart failure; ⑫ Patients with blood uric acid > 480 μmol/L and combined with any of the following: uric acid nephrolithiasis or renal function impairment (eGFR ≤ 89 ml/(min·1.73 m²)), hypertension, impaired glucose tolerance or diabetes, dyslipidemia (any of the four lipid indicators exceeding the normal reference range), obesity (BMI ≥ 28 kg/m²), coronary heart disease, stroke, heart failure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
uric acid levels in umol/L | From enrollment to the end of treatment at 12 weeks
  Uric acid levels were measured by blood samples at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.

SECONDARY OUTCOMES:
Xanthine oxidase activity in ng/mL | From enrollment to the end of treatment at 12 weeks
  Xanthine oxidase activity was measured by blood samples at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
erythrocyte sedimentation rate in mm/h | From enrollment to the end of treatment at 12 weeks
  Erythrocyte sedimentation rates were measured by blood samples at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
antinuclear antibody in semi-quantitative | From enrollment to the end of treatment at 12 weeks
  Antinuclear antibodies were measured by blood samples at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
blood glucose in mmol/L | From enrollment to the end of treatment at 12 weeks
  Blood glucoses were measured by blood samples at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
total cholesterol in mmol/L | From enrollment to the end of treatment at 12 weeks
  Total cholesterols were measured by blood samples at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
triglycerides in mmol/L | From enrollment to the end of treatment at 12 weeks
  Triglycerides were measured by blood samples at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
high-density lipoprotein cholesterol in mmol/L | From enrollment to the end of treatment at 12 weeks
  High-density lipoprotein cholesterols were measured by blood samples at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
low-density lipoprotein cholesterol in mmol/L | From enrollment to the end of treatment at 12 weeks
  Low-density lipoprotein cholesterols were measured by blood samples at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
C-reactive protein in mg/L | From enrollment to the end of treatment at 12 weeks
  C-reactive proteins were measured by blood samples at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
white blood cell count in 10^9/L | From enrollment to the end of treatment at 12 weeks
  White blood cell counts were measured by blood samples at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
leptin level in pg/mL | From enrollment to the end of treatment at 12 weeks
  Leptin levels were measured by blood samples at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
adiponectin level in ug/mL | From enrollment to the end of treatment at 12 weeks
  Adiponectin levels were measured by blood samples at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
IL-1β in pg/mL | From enrollment to the end of treatment at 12 weeks
  IL-1β levels were measured by blood samples at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
IL-2 in pg/mL | From enrollment to the end of treatment at 12 weeks
  IL-2 levels were measured by blood samples at two time points: the day of enrollment and 12 weeks after enrollment.
IL-4 in pg/mL | From enrollment to the end of treatment at 12 weeks
  IL-4 levels were measured by blood samples at two time points: the day of enrollment and 12 weeks after enrollment.
IL-6 in pg/mL | From enrollment to the end of treatment at 12 weeks
  IL-6 levels were measured by blood samples at two time points: the day of enrollment and 12 weeks after enrollment.
IL-10 in pg/mL | From enrollment to the end of treatment at 12 weeks
  IL-10 levels were measured by blood samples at two time points: the day of enrollment and 12 weeks after enrollment.
IFN-γ in pg/mL | From enrollment to the end of treatment at 12 weeks
  IFN-γ levels were measured by blood samples at two time points: the day of enrollment and 12 weeks after enrollment.
TNF-α in pg/mL | From enrollment to the end of treatment at 12 weeks
  TNF-α levels were measured by blood samples at two time points: the day of enrollment and 12 weeks after enrollment.
height in centimeters | From enrollment to the end of treatment at 12 weeks
  Height in centimeters were measured by Manual Height Ruler at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
weight in kilograms | From enrollment to the end of treatment at 12 weeks
  Weight in kilograms were measured by the Inbody 770 instrument at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
BMI in kg/m^2 | From enrollment to the end of treatment at 12 weeks
  Weight and height will be combined to report BMI in kg/m^2 at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
body fat rate in % | From enrollment to the end of treatment at 12 weeks
  Body fat rates were measured by the Inbody 770 instrument at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
muscle mass in kilograms | From enrollment to the end of treatment at 12 weeks
  Muscle masses were measured by were measured by the Inbody 770 instrument at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
basal metabolic rate in kcal | From enrollment to the end of treatment at 12 weeks
  Basal metabolic rates were measured by the Inbody 770 instrument at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
skeletal muscle mass in kilograms | From enrollment to the end of treatment at 12 weeks
  Skeletal muscle masses were measured by the Inbody 770 instrument at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
blood pressure in mmHg | From enrollment to the end of treatment at 12 weeks
  Blood pressures were measured by electronic blood pressure monitor at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
waist circumference in millimeters | From enrollment to the end of treatment at 12 weeks
  Waist circumferences were measured by tape measure at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
hip circumference in millimeters | From enrollment to the end of treatment at 12 weeks
  Hip circumferences were measured by tape measure at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
upper arm circumference in millimeters | From enrollment to the end of treatment at 12 weeks
  Upper arm circumferences were measured by tape measure at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
left hand grip strength in pound-force | From enrollment to the end of treatment at 12 weeks
  Left hand grip strengths were measured by grip dynamometer at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
right hand grip strength in pound-force | From enrollment to the end of treatment at 12 weeks
  Right hand grip strengths were measured by grip dynamometer at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
triceps skinfold thickness in millimeters | From enrollment to the end of treatment at 12 weeks
  Triceps skinfold thicknesses were measured by skin fold thickness gauge at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
subscapular horn skinfold thickness in millimeters | From enrollment to the end of treatment at 12 weeks
  Subscapular horn skinfold thicknesses were measured by skin fold thickness gauge at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
abdominal skinfold thickness in millimeters | From enrollment to the end of treatment at 12 weeks
  Abdominal skinfold thicknesses were measured by skin fold thickness gauge at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.
food intake dose in grams | From enrollment to the end of treatment at 12 weeks
  Data of food intake doses were taken by food frequency questionnaire and 3-day food diary at four time points: the day of enrollment, 4 weeks after enrollment, 8 weeks after enrollment and 12 weeks after enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Xicheng District, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cui M, Shao L, Zhao S, Guo Q, Liu X, Liu P. Effects of barley green on uric acid, inflammatory factors, xanthine oxidase activity and body composition of patients with hyperuricemia: a randomized controlled trial. Front Nutr. 2025 Oct 31;12:1684829. doi: 10.3389/fnut.2025.1684829. eCollection 2025. PMID 41245398